CLINICAL TRIAL: NCT05340049
Title: Early Craniosacral Therapy Improves Infant Neurodevelopment in Apparently Healthy Children.
Brief Title: Craniosacral Therapy Improves Infant Neurodevelopment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Gema Leon (Other)
Responsible Party: Principal Investigator, GEMA LEÓN BRAVO, Principal Investigator, Clinica Gema Leon
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ART-GLB-TTO RPA Y BC
Record Dates: First submitted 2021-12-18; First posted 2022-04-21 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Child Development Disorder
Keywords: Craniosacral treatment; primitive reflexes; cranial blocks; childhood; physiotherapy
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Intervention Model Description: 120 pupils aged 3-8 years were divided into four treatment groups set as follows: Placebo craniosacral group (n=30) Rhythmic Movement Therapy Group (n=30) Placebo of Rhythmic Movement Therapy Group (n=30) Craniosacral Therapy Group (n=30) Such participants were included according to the number of Active Primitive Reflexes (Moro, asymmetric and symmetric cervical) and/or Cranial Blocks (swaying of the dura mater, sphenoid bone and cranial parietal areas) presented by each of them
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Primary Group "Placebo of craniosacral therapy" (Placebo Comparator): 30 patients of the total sample are part of one of the the placebo group, being these patients active primitive reflexes and/or cranial blocks in smaller quantities than the other participants of the study.
  The hands were placed imitating craniosacral techinques without having any type of benefit.
  Interventions: Procedure: Academic behavioral intervention of teachers; Procedure: Therapy sessions
- Tertiary group "Rhythmic Movement Therapy" (Active Comparator): 30 patients of the total sample are part of the rhythmic movement therapy group, having 1 or all of the primitive reflexes active and/or cranial blocks studied. Exercises were applied to inhibit primitive reflex
  Interventions: Procedure: Academic behavioral intervention of teachers; Procedure: Therapy sessions
- Quaternary group "Craniosacral Therapy" (Experimental): 30 patients of the total sample are part of the rhythmic movement therapy group, having 1 or all of the primitive reflexes active and/or cranial blocks studied. Craniosacral tecniques were applied to eliminate cranial blocks and inhibit primitive reflexes
  Interventions: Procedure: Academic behavioral intervention of teachers; Procedure: Therapy sessions
- Secondary group "Placebo of Rhythmic Movement Therapy" (Placebo Comparator): 30 patients of the total sample are part of one of the the placebo group, being these patients without active primitive reflexes and/or cranial blocks, or in smaller quantities than the other participants of the study. Exercise were applied that pretend to inhibit primitive reflex, but there is no benefit
  Interventions: Procedure: Academic behavioral intervention of teachers; Procedure: Therapy sessions

INTERVENTIONS:
Procedure: Academic behavioral intervention of teachers — the school teachers examined neurobehavioral aspects of the students using the "Battelle Developmental Inventory" (BDI), which evaluates five areas of development (personal/social, adaptive, motor, communicative and cognitive) between 2 and 8 years of age. Evaluation of the Battelle scale was carried out before and after the therapy sessions.
Procedure: Therapy sessions — Seven sessions were given to each of the three groups according to their classification (PCST, PMRT, TMR, TCS), being able to obtain a stable value in each of the treatments carried out. Before each session, the effect of the previous session was explored in order to evaluate its efficacy (from the second session onwards). Each of the therapies had the same number of sessions (1 per week for 7 weeks) in order to have equality in all the parameters evaluated.
  The effectiveness values of the cranial blocks and primitive reflexs therapies were expressed as block or normal and active or inactive, depending on what finds the physiotherapist in his evaluation

SUMMARY:
Craniosacral exploration and therapy is one of the innovative palpation and treatment techniques in specialized physiotherapy, which can contribute in an efficient, subtle and sudden way to the detection of dysfunctions in the cranial sutures or fontanelles and/or alterations or blockages that may exist in the frontal lobes and other areas of the skull and body. Objective: To compare the effectiveness of craniosacral therapy with respect to traditional primitive reflex treatment therapy and how it influences the neurodevelopment of the healthy child through the Battelle scale, and to test the effectiveness of both therapies witn their placebos. Methodology: 120 children were treated without excluding sex divided into four groups: placebo group of craniosacral therapy (n=30), Placebo group of rythmic Movement Therapy (n=30), rhytmic movement therapy (n=30) and craniosacral therapy group (n=30).

DETAILED DESCRIPTION:
The growth of the individual is linked to differentiated medical-scientific stages. Physiology stipulates stages in the development and maturation of the human being, from the moment of fertilization until the day of death, due to the existence of relatively similar patterns in all human beings, produced at specific parallel times.

Primitive Reflexes (PR) are one of the patterns that are activated from the moment of birth and remain until a maximum time of 3 years of age. After this period of time, alterations in the Central Nervous System (CNS) are usually considered possible when they persist, inhibiting the maturation of motor neurons causing postural reflexes (coming from PR) to be delayed in their appearance or not to be adequately presented, including the possibility of their complete absence.

Child neurology affirms that cortical and spinal control in the newborn (NB) motor system should be the basis for the opening to higher level functions required by the growth and maturation of the CNS. The participation of the frontal lobes is essential in the rapidity of response to a stimulus, since they direct the planning of complex activities, their final conceptualization and the sustained modification of the components to arrive at an efficient motor sequence. In such a way that the frontal lobes provide a kind of synergism with the rest of the CNS, promoting a faster impulse to think, speak and act. That is why, when there is a lesion in such areas, it can cause the reduction of such impulses and generate deterioration and/or delays at neurobehavioral and neuropsychological levels. The cranial sutures or fontanelles are dense fibrous bands that serve as interconnections of the cranial bones. They are critical in the NB, as during delivery they allow the head to pass through the vaginal canal without putting pressure on the baby's brain. After delivery, the sutures remain open for several months of life for the development, growth and protection of the brain. Palpation of the cranial sutures or fontanelles is one of the practices in neurology and physical therapy used to determine the growth and development of the child.

Craniosacral exploration and therapy is one of the innovative palpation and treatment techniques in specialized physical therapy, which can contribute in an efficient, subtle and sudden way to the detection of dysfunctions in the cranial sutures or fontanelles and/or in the alterations or blockages that may exist in the frontal lobes and other areas of the skull and body. The manual skill of craniosacral exploration is based on the ability of the craniosacral therapist to feel the state of the fasciae surrounding the brain and spinal cord, as well as their physiological structure. The gentle, non-invasive manual contact, with hardly any pressure, contributes to the detection of tensions in the connective tissue, which could lead to possible disruptions in the treated patient. This is how the specialized therapist assesses the rhythm of mobility of the cranial fasciae, their synchrony, strength, frequency and tenacity. When there are alterations in the structure and state of the cranial membranes diagnosed by the specialized therapist, craniosacral therapy would be initiated to balance the membrane tensions of the bones that make up the skull and normalize the movement, synchrony, strength, frequency and tenacity. Failure to release the existing tensions in the fascial system could lead to different imbalances in the nervous, visceral, endocrine and circulatory systems, both blood and lymphatic; this could cause states of persistent RP or its reactivation, cranial blockages that do not allow the correct neurological and cognitive functioning, and possible mental and learning disorders or alterations.

The studies that have been carried out in Physiotherapy at behavioral and neuropsychological level show that there is a high percentage of relationship between persistent RPs and certain disorders, such as attention deficit, hyperactivity, depression, autism and poor concentration, but such dysfunctions are not only described in children with clear pathologies such as those mentioned above, but studies have also been presented in the child population characterized as healthy, with mild patterns of alterations in their cognitive, motor, psychological and social development that show different degrees of activation of RPs. Therefore, it is necessary to evaluate all stages of child development (from gestation to the onset of puberty) to obtain a complete neurological chronological assessment. Other studies show that tensions in the temporo-mandibular joints, in the frontal and parietal areas of the skull, cause problems such as migraines, delayed motor behavior, stress, anxiety, bruxism and lack of concentration, leading to different disorders that occur as the condition progresses, helping to worsen the physical and mental well-being of the child. Thus, craniosacral therapy indicates that all these disorders mentioned in healthy children may be due to a plastic deformation in any of the cranial membranes, which, when generalized to the rest of the body, may influence the degree of fascial tension of the others. With the restructuring of these fasciae by means of craniosacral therapy, the integrity of the organism and thus its well-being would return.

This work is based on the previous research presented as Master's Thesis under the name of "Early Craniosacral and Primitive Reflex Evaluation in Child Neurodevelopment" by Leon et al (2020). Where 14 PR and 6 BC were assessed in a group of 120 children divided into two age ranges: 3 to 5 and 6 to 8 years old, resulting in the following conclusions:

1. Those considered as gestation and/or complicated deliveries suppose risk factors for the active presence of primitive reflexes and existence of craniocranial blocks.
2. The frequency of activation of the primitive reflexes of Moro and cervical symmetric, increases with age (in the studied range) without relation to gender, a result in contrast to that expected according to the normal development of the infant.
3. When the neurodevelopmental assessment measured according to the Battelle scale is shown in low (0-50%) or high (80-100%) ranges, the frequency of activation of the asymmetric and symmetric cervical reflexes and of blocks of the sphenoid bone, dura mater rocking and parietal bones is higher, ordered according to the degree of frequency.
4. The presence of certain activated primitive reflexes (Moro reflex and cervical asymmetric and symmetric) is significantly related to blockages of some areas of the craniosacral system (swaying of the dura mater and sphenoid bone).

The main objective of this work is to to compare the effectiveness of craniosacral therapy with respect to traditional primitive reflex treatment therapy and how it influences the neurodevelopment of the healthy child through the Battelle scale, and to test the effectiveness of both therapies witn their placebos.

Thus, our aims are to compare the effectiveness of craniosacral therapy with respect to traditional primitive reflex treatment therapy and how it influences the neurodevelopment of the apparently healthy child through the Battelle scale, as well as to examine which of the two therapies would be faster in inhibiting RPA and to test the effectiveness of both therapies witn their respect placebos

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy children
* School group
* Within age range

Exclusion Criteria:

* Children with possible pathologies
* Older than the established age

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2021-12-18 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Previous teachers' test by means of the "Battelle Development Inventory" (BDI). | five months
  The school teachers examined neurobehavioral aspects of the students using the "Battelle Developmental Inventory" (BDI), which assesses five areas of development (personal/social, adaptive, motor, communicative and cognitive) between 2 and 8 years of age. The results are assigned in age-adjusted percentages, classified as: low (0-50%), normal (50-80%) and high (80-100%). Low and high values are considered impairments in one or more of the evaluated areas.
  The minimum and maximum values are 0-341. 170.5-272.8 in item scores are ideal values that indicate normal behavior according to their age.

SECONDARY OUTCOMES:
Presence of active primitive reflex and cranial blocks | two months
  physical examination measure the presence of APR and CB by an experienced physiotherapist

CONTACTS AND LOCATIONS:
Overall Officials: Irene Cantarero Carmona, Study chair, Study Chair — Universidad de Córdoba
Locations (1):
- Gema León Physiotherapy and Rehabilitation Clinic, Córdoba, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No
: No The request for data will be studied and considered upon justified request.

REFERENCES:
- [Background] Tomassini A, Spinelli D, Jacono M, Sandini G, Morrone MC. Rhythmic oscillations of visual contrast sensitivity synchronized with action. J Neurosci. 2015 May 6;35(18):7019-29. doi: 10.1523/JNEUROSCI.4568-14.2015. PMID 25948254
- [Background] Schaffert N, Janzen TB, Mattes K, Thaut MH. A Review on the Relationship Between Sound and Movement in Sports and Rehabilitation. Front Psychol. 2019 Feb 12;10:244. doi: 10.3389/fpsyg.2019.00244. eCollection 2019. PMID 30809175
- [Background] Ortiz-Campoy S, Lirio-Romero C, Romay-Barrero H, Alvarez DM, Lopez-Munoz P, Palomo-Carrion R. The Role of Physiotherapy in Pediatric Palliative Care: A Systematic Review. Children (Basel). 2021 Nov 12;8(11):1043. doi: 10.3390/children8111043. PMID 34828756
- [Background] Larsson I, Miller M, Liljedahl K, Gard G. Physiotherapists' experiences of physiotherapy interventions in scientific physiotherapy publications focusing on interventions for children with cerebral palsy: a qualitative phenomenographic approach. BMC Pediatr. 2012 Jul 2;12:90. doi: 10.1186/1471-2431-12-90. PMID 22747596
- [Background] Lucas BR, Elliott EJ, Coggan S, Pinto RZ, Jirikowic T, McCoy SW, Latimer J. Interventions to improve gross motor performance in children with neurodevelopmental disorders: a meta-analysis. BMC Pediatr. 2016 Nov 29;16(1):193. doi: 10.1186/s12887-016-0731-6. PMID 27899082
- [Background] Das SP, Ganesh GS. Evidence-based Approach to Physical Therapy in Cerebral Palsy. Indian J Orthop. 2019 Jan-Feb;53(1):20-34. doi: 10.4103/ortho.IJOrtho_241_17. PMID 30905979
- [Background] Degerstedt F, Wiklund M, Enberg B. Physiotherapeutic interventions and physical activity for children in Northern Sweden with cerebral palsy: a register study from equity and gender perspectives. Glob Health Action. 2016 Jan-Dec;10(sup2):1272236. doi: 10.1080/16549716.2017.1272236. PMID 28219314
- [Background] Hartley H, Cassidy E, Bunn L, Kumar R, Pizer B, Lane S, Carter B. Exercise and Physical Therapy Interventions for Children with Ataxia: A Systematic Review. Cerebellum. 2019 Oct;18(5):951-968. doi: 10.1007/s12311-019-01063-z. PMID 31392562
- [Background] Gonzalez-Santos J, Gonzalez-Bernal JJ, De-la-Fuente Anuncibay R, Soto-Camara R, Cubo E, Aguilar-Parra JM, Trigueros R, Lopez-Liria R. Infant Cranial Deformity: Cranial Helmet Therapy or Physiotherapy? Int J Environ Res Public Health. 2020 Apr 10;17(7):2612. doi: 10.3390/ijerph17072612. PMID 32290217
- [Background] Ryan JM, Cassidy EE, Noorduyn SG, O'Connell NE. Exercise interventions for cerebral palsy. Cochrane Database Syst Rev. 2017 Jun 11;6(6):CD011660. doi: 10.1002/14651858.CD011660.pub2. PMID 28602046
- [Background] Sinha AG, Sharma R. Factors Influencing Utilization of Physiotherapy Service among Children with Cerebral Palsy in Jalandhar District of Punjab. J Neurosci Rural Pract. 2017 Apr-Jun;8(2):209-215. doi: 10.4103/0976-3147.203852. PMID 28479794
- [Background] Okenwa W, Edeh A. A review of clinical presentation and physiotherapy management of cerebral palsy patients in Esut teaching hospital, Enugu, Nigeria. Afr Health Sci. 2019 Dec;19(4):3085-3090. doi: 10.4314/ahs.v19i4.30. PMID 32127884
- [Background] Nielsen G, Stone J, Matthews A, Brown M, Sparkes C, Farmer R, Masterton L, Duncan L, Winters A, Daniell L, Lumsden C, Carson A, David AS, Edwards M. Physiotherapy for functional motor disorders: a consensus recommendation. J Neurol Neurosurg Psychiatry. 2015 Oct;86(10):1113-9. doi: 10.1136/jnnp-2014-309255. Epub 2014 Nov 28. PMID 25433033
- [Background] Pecuch A, Gieysztor E, Telenga M, Wolanska E, Kowal M, Paprocka-Borowicz M. Primitive Reflex Activity in Relation to the Sensory Profile in Healthy Preschool Children. Int J Environ Res Public Health. 2020 Nov 6;17(21):8210. doi: 10.3390/ijerph17218210. PMID 33172138
- [Background] Gieysztor EZ, Choinska AM, Paprocka-Borowicz M. Persistence of primitive reflexes and associated motor problems in healthy preschool children. Arch Med Sci. 2018 Jan;14(1):167-173. doi: 10.5114/aoms.2016.60503. Epub 2016 Jun 13. PMID 29379547
- [Background] Bob P, Konicarova J, Raboch J. Disinhibition of Primitive Reflexes in Attention Deficit and Hyperactivity Disorder: Insight Into Specific Mechanisms in Girls and Boys. Front Psychiatry. 2021 Nov 8;12:430685. doi: 10.3389/fpsyt.2021.430685. eCollection 2021. PMID 34819879
- [Background] Konicarova J, Bob P, Raboch J. Persisting primitive reflexes in medication-naive girls with attention-deficit and hyperactivity disorder. Neuropsychiatr Dis Treat. 2013;9:1457-61. doi: 10.2147/NDT.S49343. Epub 2013 Sep 20. PMID 24092983
- [Background] Melillo R, Leisman G, Mualem R, Ornai A, Carmeli E. Persistent Childhood Primitive Reflex Reduction Effects on Cognitive, Sensorimotor, and Academic Performance in ADHD. Front Public Health. 2020 Nov 17;8:431835. doi: 10.3389/fpubh.2020.431835. eCollection 2020. PMID 33282806
- [Background] Nguyen AT, Armstrong EA, Yager JY. Neurodevelopmental Reflex Testing in Neonatal Rat Pups. J Vis Exp. 2017 Apr 24;(122):55261. doi: 10.3791/55261. PMID 28518104
- [Background] Sohn M, Ahn Y, Lee S. Assessment of Primitive Reflexes in High-risk Newborns. J Clin Med Res. 2011 Dec;3(6):285-90. doi: 10.4021/jocmr706w. Epub 2011 Nov 10. PMID 22393339
- [Background] Marin Gabriel MA, Olza Fernandez I, Malalana Martinez AM, Gonzalez Armengod C, Costarelli V, Millan Santos I, Fernandez-Canadas Morillo A, Perez Riveiro P, Lopez Sanchez F, Garcia Murillo L. Intrapartum synthetic oxytocin reduce the expression of primitive reflexes associated with breastfeeding. Breastfeed Med. 2015 May;10(4):209-13. doi: 10.1089/bfm.2014.0156. Epub 2015 Mar 18. PMID 25785487
- [Background] Futagi Y, Toribe Y, Suzuki Y. The grasp reflex and moro reflex in infants: hierarchy of primitive reflex responses. Int J Pediatr. 2012;2012:191562. doi: 10.1155/2012/191562. Epub 2012 Jun 11. PMID 22778756
- [Background] Gieysztor E, Pecuch A, Kowal M, Borowicz W, Paprocka-Borowicz M. Pelvic Symmetry Is Influenced by Asymmetrical Tonic Neck Reflex during Young Children's Gait. Int J Environ Res Public Health. 2020 Jul 2;17(13):4759. doi: 10.3390/ijerph17134759. PMID 32630679
- [Background] Huber SJ, Paulson GW. Relationship between primitive reflexes and severity in Parkinson's disease. J Neurol Neurosurg Psychiatry. 1986 Nov;49(11):1298-300. doi: 10.1136/jnnp.49.11.1298. PMID 3794736
- [Background] Haller H, Lauche R, Cramer H, Rampp T, Saha FJ, Ostermann T, Dobos G. Craniosacral Therapy for the Treatment of Chronic Neck Pain: A Randomized Sham-controlled Trial. Clin J Pain. 2016 May;32(5):441-9. doi: 10.1097/AJP.0000000000000290. PMID 26340656
- [Background] Curtis P, Gaylord SA, Park J, Faurot KR, Coble R, Suchindran C, Coeytaux RR, Wilkinson L, Mann JD. Credibility of low-strength static magnet therapy as an attention control intervention for a randomized controlled study of CranioSacral therapy for migraine headaches. J Altern Complement Med. 2011 Aug;17(8):711-21. doi: 10.1089/acm.2010.0277. Epub 2011 Jul 6. PMID 21732734
- [Background] Mann JD, Faurot KR, Wilkinson L, Curtis P, Coeytaux RR, Suchindran C, Gaylord SA. Craniosacral therapy for migraine: protocol development for an exploratory controlled clinical trial. BMC Complement Altern Med. 2008 Jun 9;8:28. doi: 10.1186/1472-6882-8-28. PMID 18541041
- [Background] Haller H, Lauche R, Sundberg T, Dobos G, Cramer H. Craniosacral therapy for chronic pain: a systematic review and meta-analysis of randomized controlled trials. BMC Musculoskelet Disord. 2019 Dec 31;21(1):1. doi: 10.1186/s12891-019-3017-y. PMID 31892357
- [Background] Mataran-Penarrocha GA, Castro-Sanchez AM, Garcia GC, Moreno-Lorenzo C, Carreno TP, Zafra MD. Influence of craniosacral therapy on anxiety, depression and quality of life in patients with fibromyalgia. Evid Based Complement Alternat Med. 2011;2011:178769. doi: 10.1093/ecam/nep125. Epub 2011 Jun 15. PMID 19729492
- [Background] Parnell Prevost C, Gleberzon B, Carleo B, Anderson K, Cark M, Pohlman KA. Manual therapy for the pediatric population: a systematic review. BMC Complement Altern Med. 2019 Mar 13;19(1):60. doi: 10.1186/s12906-019-2447-2. PMID 30866915
- [Background] Golanska P, Saczuk K, Domarecka M, Kuc J, Lukomska-Szymanska M. Temporomandibular Myofascial Pain Syndrome-Aetiology and Biopsychosocial Modulation. A Narrative Review. Int J Environ Res Public Health. 2021 Jul 23;18(15):7807. doi: 10.3390/ijerph18157807. PMID 34360099
- [Background] Levy SE, Hyman SL. Complementary and alternative medicine treatments for children with autism spectrum disorders. Child Adolesc Psychiatr Clin N Am. 2008 Oct;17(4):803-20, ix. doi: 10.1016/j.chc.2008.06.004. PMID 18775371
- [Background] Guillaud A, Darbois N, Monvoisin R, Pinsault N. Reliability of Diagnosis and Clinical Efficacy of Cranial Osteopathy: A Systematic Review. PLoS One. 2016 Dec 9;11(12):e0167823. doi: 10.1371/journal.pone.0167823. eCollection 2016. PMID 27936211
- [Background] Park Y, Kabariti J, Tafler L. Craniosacral Therapy Use in Normal Pressure Hydrocephalus. Cureus. 2021 May 7;13(5):e14886. doi: 10.7759/cureus.14886. PMID 34109075
- [Background] Wittman RA, Vallone SA. Inclusion of chiropractic care in multidisciplinary management of a child with Prader-Willi syndrome: a case report. J Chiropr Med. 2009 Dec;8(4):193-9. doi: 10.1016/j.jcm.2009.08.001. PMID 19948310
- [Background] Kuc J, Szarejko KD, Golebiewska M. Evaluation of Soft Tissue Mobilization in Patients with Temporomandibular Disorder-Myofascial Pain with Referral. Int J Environ Res Public Health. 2020 Dec 21;17(24):9576. doi: 10.3390/ijerph17249576. PMID 33371343
- [Background] Adragna V, Bertino AS, Carano M, Soru A, Taranto G, Desideri R. O052. Migraine without aura and osteopathic medicine, a non-pharmacological approach to pain and quality of life: open pilot study. J Headache Pain. 2015 Dec;16(Suppl 1):A180. doi: 10.1186/1129-2377-16-S1-A180. No abstract available. PMID 28132208
- [Background] Do TP, Heldarskard GF, Kolding LT, Hvedstrup J, Schytz HW. Myofascial trigger points in migraine and tension-type headache. J Headache Pain. 2018 Sep 10;19(1):84. doi: 10.1186/s10194-018-0913-8. PMID 30203398